CLINICAL TRIAL: NCT03752905
Title: A Phase 1/2 Randomized, Saline-Controlled, Single-Blind, Multiple Ascending Dose, Dose-Escalation, Multi-Center Trial of PTR-01 in Adult Patients With Recessive Dystrophic Epidermolysis Bullosa (RDEB)
Brief Title: A Phase 1/2 Trial of PTR-01 in Adult Patients With Recessive Dystrophic Epidermolysis Bullosa (RDEB)
Acronym: PTR-01-001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Phoenix Tissue Repair, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTR-01-001
Record Dates: First submitted 2018-11-19; First posted 2018-11-26 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Recessive Dystrophic Epidermolysis Bullosa
Keywords: RDEB
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, Saline-Controlled, Single-Blind, Multiple Ascending Dose, Dose-Escalation, Multi-Center
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PTR-01 0.1 mg/kg (Experimental): Three intravenous infusions of PTR-01 at 0.1 mg/kg with doses 2 weeks apart.
  Interventions: Drug: PTR-01
- PTR-01 0.3 mg/kg (Experimental): Three intravenous infusions of PTR-01 at 0.3 mg/kg with doses 2 weeks apart.
  Interventions: Drug: PTR-01
- PTR-01 1.0 mg/kg (Experimental): Three intravenous infusions of PTR-01 at 1.0 mg/kg with doses 2 weeks apart.
  Interventions: Drug: PTR-01
- Normal Saline (Placebo Comparator): Saline control to mimic PTR-01.
  Interventions: Drug: Normal saline
- PTR-01 3.0 mg/kg (Experimental): Three intravenous infusions of PTR-01 at 3.0 mg/kg with doses 2 weeks apart.
  Interventions: Drug: PTR-01

INTERVENTIONS:
Drug: PTR-01 — Recombinant human collagen 7 (rC7)
  Other Names: Recombinant human collagen 7 (rC7)
  Arms: PTR-01 0.1 mg/kg; PTR-01 0.3 mg/kg; PTR-01 1.0 mg/kg; PTR-01 3.0 mg/kg
Drug: Normal saline — Saline control
  Arms: Normal Saline

SUMMARY:
Protocol PTR-01-001 is a Phase 1/2 study of PTR-01.

The study is divided into an up to 4-week Screening Period, a 10-week Treatment Period and an 8-week Follow-up Period.

Cohorts 1, 2, 3 and 4 will consist of 2, 4, 3 and 3 patients respectively. Each cohort will consist of patients divided into two groups (Group 1 and Group 2) randomized in a 1:1 ratio. Patients in Group 1 will receive three doses of active drug followed by 3 doses of saline control. Patients in Group 2 will receive three doses of saline control followed by 3 doses of active drug.

Cohort 1 patients randomized to Group 1 will receive 3 doses of active treatment (PTR-01) at a dose of 0.1 mg/kg followed by 3 doses of saline control for a total of 6 doses. Cohort 1 patients randomized to Group 2 will receive 3 doses of saline control followed by 3 doses of active treatment (PTR-01) at a dose of 0.1 mg/kg for a total of 6 doses.

DETAILED DESCRIPTION:
Protocol PTR-01-001 is a saline-controlled, single and repeat dose, dose-escalation, crossover study designed to determine the safety, tolerability, tissue kinetics, pharmacodynamics and preliminary efficacy of PTR 01.

The study is divided into three periods: an up to 4-week Screening Period, a 10-week Treatment Period and an 8-week Follow-up Period. During the Screening Period and Follow-up Period there will be no study drug treatment.

During the Treatment Period a total of 3 doses of PTR-01 and 3 doses of saline control will be administered to patients for a total of 6 doses over a 10-week period in three cohorts dosed at 0.1, 0.3, 1.0 and 3.0 mg/kg (active drug). Twelve patients with a diagnosis of RDEB and a history of at least one chronic wound will be enrolled. Those patients who do not have documentation of genetic analysis and IF staining will have blood for genetic analysis and a biopsy for IF staining prior to enrollment (both required).

Cohorts 1, 2, 3 and 4 will consist of 2, 4, 3 and 3 patients respectively. Each cohort will consist of patients divided into two groups (Group 1 and Group 2) randomized in a 1:1 ratio. Patients will receive doses 2 weeks apart. Patients in Group 1 will receive three doses of active drug followed by 3 doses of saline control. Patients in Group 2 will receive three doses of saline control followed by 3 doses of active drug. This cross-over design will yield a total of 14 patients all of whom will receive active drug and saline control.

Prior to randomization, patients will complete a Screening Period to assess the extent and impact of skin disease involvement and the chronicity of at least one wound. Only patients who meet all of the eligibility criteria will be randomized for treatment.

Cohort 1 patients randomized to Group 1 will receive 3 doses of active treatment (PTR-01) at a dose of 0.1 mg/kg followed by 3 doses of saline control for a total of 6 doses. Cohort 1 patients randomized to Group 2 will receive 3 doses of saline control followed by 3 doses of active treatment (PTR-01) at a dose of 0.1 mg/kg for a total of 6 doses. After the last patient in Cohort 1 has received their third dose and safety labs for all patients have been reviewed by the Data Safety Monitoring Board (DSMB), the next cohort may be enrolled. This same schedule and safety review process will be followed for all subsequent dosing cohorts, with Cohort 2, Cohort 3 and Cohort 4 receiving 0.3, 1.0 and 3.0 mg/kg respectively.

Efficacy assessments will be performed prior to first dose of therapy (at the end of the Screening Period), after the last dose of study drug in Period 1, after the last dose of study drug in Period 2 of the Treatment Period and 2 weeks (Day 85) after the last dose of study drug (at the end of the Follow-up Period).

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 16 years of age.
2. Has signed the current approved informed consent form.
3. Has a diagnosis of RDEB based on genetic analysis and consistent with a recessive inheritance pattern.
4. Has deficient C7 staining at the dermal-epidermal junction (DEJ) by IF.
5. Has at least 1 unhealed wound 10-200 cm2 for at least 6 weeks at the Screening Visit.
6. Agrees to use contraception as follows:

   * For women of childbearing potential (WOCBP) agrees to use highly effective contraceptive (including abstinence) methods from Screening, through the study, and for at least 10 weeks after the last dose of study drug. Non-childbearing potential is defined as a female who meets either of the following criteria: age ≥50 years and no menses for at least 1 year or documented hysterectomy, bilateral tubal ligation, or bilateral oophorectomy (see Section 7.4.1.2 for details on the definition of non-childbearing potential).
   * For males, agrees to use a condom with any WOCBP sexual partner from Day 1 of study treatment, through the study, and at least 10 weeks after the last dose of study drug.
7. Be willing and able to comply with this protocol.

Exclusion Criteria:

1. Has known systemic hypersensitivity to any of the inactive ingredients in PTR-01.
2. Is pregnant or nursing.
3. Has received in the last six months any investigational gene therapy product or in the last three months any non-gene therapy investigational products.
4. Is anticipated to receive new regimens of antibiotics or other anti-infectives during the trial.
5. Has any other medical or personal condition that, in the opinion of the Investigator, may potentially compromise the safety or compliance of the patient, or may preclude the patient's successful completion of the clinical study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Up to Day 127
  The primary endpoint of this study is safety and tolerability, as assessed by treatment-emergent adverse events, infusion-associated reactions (IAR) and immunogenicity

SECONDARY OUTCOMES:
To measure the peak serum concentration (Cmax) of PTR-01 | Pre-dose, 15 minutes, 60 minutes, 2 hours, 4 hours, 8 hours and 24 hours post-dose
  Pharmacokinetic parameter estimates of Cmax
To measure the time to peak concentration (Tmax) of PTR-01 | Pre-dose, 15 minutes, 60 minutes, 2 hours, 4 hours, 8 hours and 24 hours post-dose
  Pharmacokinetic parameter estimates of Tmax
To measure the area under the curve (AUC) of PTR-01 | Pre-dose, 15 minutes, 60 minutes, 2 hours, 4 hours, 8 hours and 24 hours post-dose
  Pharmacokinetic parameter estimates of AUC
To measure the clearance of PTR-01 | Pre-dose, 15 minutes, 60 minutes, 2 hours, 4 hours, 8 hours and 24 hours post-dose
  Pharmacokinetic parameter estimates of clearance
To measure the half-life (t1/2) of PTR-01 | Pre-dose, 15 minutes, 60 minutes, 2 hours, 4 hours, 8 hours and 24 hours post-dose
  Pharmacokinetic parameter estimates of t1/2
Change from Baseline in rC7 | Screening and Day 127
  Change in rC7 on skin biopsy by immunofluorescence (IF)
Change from Baseline in anchoring fibrils | Screening and Day 127
  Change in anchoring fibrils on skin biopsy by electron microscopy (EM)
Duration of rC7 residence in tissue | Screening and Day 127
  Duration of rC7 residence in tissue by skin biopsy

OTHER OUTCOMES:
Change from Baseline in suction blister time | Baseline and Day 127
  Change from Baseline in suction blister time (as compared to placebo and historical controls)
Change from Baseline in target wound size | Baseline and Day 127
  Change from Baseline in target wound size (percent healing from Baseline)
Change from Baseline in healing of up to 5 chronic wounds | Baseline and Day 127
  Change in healing of up to 5 wounds that chronically heal and reopen
Change from Baseline in wound surface area | Screening and Day 127
  Change from Baseline in wound surface area
Change from Baseline in patient reported outcomes as assessed by the Leuven Itch Scale (LIS) | Baseline and Day 127
  Change from Baseline in patient reported outcomes
Change from Baseline in patient reported outcomes as assessed by the pruritus-specific quality-of-life instrument ("ItchyQoL") | Baseline and Day 127
  Change from Baseline in patient reported outcomes
Change from Baseline in patient reported outcomes as assessed by the Quality of Life in Epidermolysis Bullosa (QOLEB) Questionnaire | Baseline and Day 127
  Change from Baseline in patient reported outcomes
Change from Baseline in patient reported outcomes as assessed by the full Health Assessment Questionnaire (HAQ) | Baseline and Day 127
  Change from Baseline in patient reported outcomes
Change from Baseline in the Investigator Global Assessment | Screening and Day 127
  Change from Baseline in the Investigator Global Assessment (IGA)
Change from Baseline in the biochemical marker albumin | Screening and Day 127
  Change from Baseline in biochemical markers of disease (albumin)
Change from Baseline in the biochemical marker iron | Screening and Day 127
  Change from Baseline in biochemical markers of disease (iron)
Change from Baseline in the biochemical marker total iron binding capacity | Screening and Day 127
  Change from Baseline in biochemical markers of disease (total iron binding capacity)
Change from Baseline in the biochemical marker hemoglobin | Screening and Day 127
  Change from Baseline in biochemical markers of disease (hemoglobin)
Change from Baseline in the biochemical marker hematocrit | Screening and Day 127
  Change from Baseline in biochemical markers of disease (hematocrit)
Change from Baseline in the biochemical marker total protein | Screening and Day 127
  Change from Baseline in biochemical markers of disease (total protein)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Podrebarac, MD, Study Director — Phoenix Tissue Repair
Locations (3):
- United States (3):
  - Stanford University, Redwood City, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Thomas Jefferson Univeristiy, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to share individual participant data with other researchers.

REFERENCES:
- See also: Sponsor website — http://phoenixtissuerepair.com